CLINICAL TRIAL: NCT00952250
Title: Personalized and Targeted Feedback in the ACTION-Registry-GWTG
Brief Title: Targeted Feedback Reports to Improve Acute Coronary Syndromes (ACS) Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00010526
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Acute Coronary Syndromes
Keywords: quality improvement
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Feedback Reports (Active Comparator): Conventional feedback reports
  Interventions: Behavioral: Targeted Feedback Reports
- Targeted Feedback Report (Experimental): Report designed to target areas for local hospital-specific improvement.
  Interventions: Behavioral: Targeted Feedback Report

INTERVENTIONS:
Behavioral: Targeted Feedback Reports — Sites randomized to this arm will receive specialized feedback summarizing their adherence to the guidelines and suggestions on ways to improve performance.
  Arms: Targeted Feedback Reports
Behavioral: Targeted Feedback Report — Report designed to target areas for local hospital-specific improvement
  Arms: Targeted Feedback Report

SUMMARY:
This project is designed to examine the impact of tailored feedback on site performance.

The investigators' objective is to evaluate whether a 'personalized and targeted' feedback, education and performance improvement intervention has a greater impact on adherence to recommended guidelines than standard feedback.

The investigators hypothesize that a site-specific report with centrally identified targets for improvement paired with target specific interventions will enable sites to quickly identify and prioritize salient problem areas, have ready access to an analysis of factors that underlie problems, and formulate an effective action plan. The investigators also hypothesize that those hospitals randomized to receive intervention will be more likely to improve their overall performance, as well as their target specific performance, during the period of observation in direct response to activated QI processes.

Outcomes:

The primary outcome is improvement in the overall composite of all metrics eligible for intervention regardless of their selection as targets.

The secondary outcome is improvement in the composite of targeted metrics.

Outcomes will be assessed in all participating sites, and in among relevant performance subgroups (low performers, academic centers, full service, and among medication versus process metrics).

ELIGIBILITY:
Inclusion Criteria:

* hospitals participating in the ACTION Registry GWTG

Exclusion Criteria:

* sites with low volume of data submission (< 10 data forms in the past year)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is improvement in the overall composite of all metrics eligible for intervention regardless of their selection as targets. | 12 months

SECONDARY OUTCOMES:
The secondary outcome is improvement in the composite of targeted metrics. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen P Alexander, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Derived] Alexander KP, Wang TY, Li S, Lytle BL, Slattery LE, Calhoun S, Poteat J, Roe MT, Rumsfeld JS, Cannon CP, Peterson ED. Randomized trial of targeted performance feedback to facilitate quality improvement in acute myocardial infarction care. Circ Cardiovasc Qual Outcomes. 2011 Jan 1;4(1):129-35. doi: 10.1161/CIRCOUTCOMES.110.958470. PMID 21245461